CLINICAL TRIAL: NCT04894149
Title: Prehabilitation and Rehabilitation for Patients With Oesophageal Cancer
Acronym: PRESO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gabriella Alexandersson von Döbeln (Other)
Responsible Party: Sponsor-Investigator, Gabriella Alexandersson von Döbeln, Principal Investigator, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21/001
Record Dates: First submitted 2021-05-04; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapy (Experimental)
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Supervised physiotherapy one hour twice weekly and 20 minutes three times weekly during 14- 17 weeks before surgery during neoadjuvant chemotherapy or chemoradiotherapy and during eight weeks after surgery (sometimes during adjuvant chemotherapy)

SUMMARY:
Patients with oesophageal cancer selected for oncological and surgical treatment with curative intent are offered supervised physiotherapy and home-based training before and after surgery.

DETAILED DESCRIPTION:
Patients with loco-regional oesophageal cancer who will receive neoadjuvant chemotherapy or chemoradiotherapy followed by surgery and sometimes adjuvant chemotherapy are eligible to be enrolled in the trial. Study treatment is supervised group training twice weekly and home-based training three times weekly during neoadjuvant treatment and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma in the oesophagus or cardia (Siewert I or II), cT1 N+ or cT2-4a any N, M0, according to the 8th version of the AJCC TNM classification.
* Assessed at a multidisciplinary conference to be suitable for curatively intended oncological and surgical treatment.
* Age > 18 years.
* Performance status ECOG 0-2.
* Patient has provided written informed consent.

Exclusion Criteria:

* Previous radiotherapy in the thorax (except for tangential field radiotherapy for breast cancer).
* Inability to understand written and spoken instructions and to comply with protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Adherence to exercise sessions. | Up to 40 weeks
  Percentage of sessions completed out of number of sessions planned
Un-planned interruptions in the prehabilitation/rehabilitation programme | Up to 40 weeks
  Percentage of patients having an unplanned interruption of ten days or more of the supervised prehabilitation/rehabilitation programme

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No